CLINICAL TRIAL: NCT02031783
Title: Glucose:Fructose Versus Glucose Carbohydrate Ingestion and Endurance Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13.09.PER
Record Dates: First submitted 2013-11-26; First posted 2014-01-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Fructose; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- mixture of glucose and fructose (Experimental): mixture of glucose and fructose
  Interventions: Dietary Supplement: glucose
- Glucose (Active Comparator): Single glucose
  Interventions: Dietary Supplement: Mixture of glucose and fructose

INTERVENTIONS:
Dietary Supplement: Mixture of glucose and fructose
  Arms: Glucose
Dietary Supplement: glucose
  Arms: mixture of glucose and fructose

SUMMARY:
The primary objective is to show that multiple transportable carbohydrate ingestion is more effective in improving endurance performance compared to single transportable carbohydrate ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 to 60 years
* A history of competitive triathlon performance (≥ 2 years)
* Participation in at least four competitive triathlon events within the past 2 years
* Be in regular training for triathlon events
* A personal best time for a standard ½ Ironman race (1.9 km swim, 90 km cycle, 21.1 km run) in the last year of either:

  * ≤ 6 h 00 min, for men aged 18-40 years
  * or ≤6 h 05 min for men aged 40-50 years
  * or ≤6 h 20 min for men aged 50-60 years
* Alternatively, if not competed in ½ Ironman in the last year, at least one standard distance triathlon (1.5 km swim, 40 km cycle, 10 km run) within the last 12 months:

  * ≤2 h 13 min, for men aged 18-40 years
  * or ≤2 h 18 min for men aged 40-50 years
  * or ≤2 h 23 min for men aged 50-60 years
* Available to compete in the ½ Ironman events and complete all study requirements
* Experienced in using carbohydrate supplementation, as gels, bars, and drinks in training/racing, specifically at rates ≥60-90g/h)
* Experience of specific formulations may include both or only multiple and single transportable carbohydrates, thus a full assessment would be made prior to recruitment to ensure balance during randomization and account for any association with the primary outcome
* Obtained his (or his legal representative's) informed consent.

Exclusion Criteria:

* Failure to meet health requirements defined in the Health Questionnaire
* Prior known fructose intolerance
* Wheat intolerance or other precluding food or packaging-related allergies
* An existing injury affecting ability to race to best ability
* A chronic injury that may affect ability to complete the races
* Unable to carry out performance assessments and questionnaires correctly
* Unable to tolerate the treatment during the familiarization sessions
* Taking medications thought to interfere with the study outcomes
* Currently participating or having participated in another clinical study during the last four weeks prior to the beginning of this study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
TIME to finish a long distance triathlon | Total time recorded at the end of the race 1 and race 2

CONTACTS AND LOCATIONS:
Locations (1):
- Massey University, Wellington, New Zealand

REFERENCES:
- [Derived] Rowlands DS, Houltham SD. Multiple-Transportable Carbohydrate Effect on Long-Distance Triathlon Performance. Med Sci Sports Exerc. 2017 Aug;49(8):1734-1744. doi: 10.1249/MSS.0000000000001278. PMID 28350714